CLINICAL TRIAL: NCT02467699
Title: Validation of a Noninvasive Navigation System for in Vivo Measurement of the Kinematics of the Knee
Brief Title: Navigation System for in Vivo Measurement of the Kinematics of the Knee
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6158
Record Dates: First submitted 2015-05-14; First posted 2015-06-10 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Knee osteoarthritis; Knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The knee prosthesis is a validated treatment for end-stage osteoarthritis, and this intervention usually provides a significant improvement in the quality of life of patients. However, a significant percentage of patients (up 30%) say disappointed with the outcome of the intervention. One hypothesis that could explain these poor results might be poor adaptation of the implants to the patient's anatomy, resulting in a non-physiological kinematics for the patient. Multiple studies try to obtain an individual adaptation of the intervention according to multiple criteria. The measurement of the kinematics of the knee before surgery could participate in this process.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients operated in the service in 2014 to care for end-stage knee osteoarthritis by implantation of a total hip knee prosthesis.

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated in the service in 2014 to care for end-stage knee osteoarthritis by implantation of a total knee prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
in vivo measurement of the kinematics of the knee | patient's medical data will be collected by health professional for the duration hospital stay, up to 1 year]

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Centre de Chirurgie Orthopédique et de la Main (CCOM), Strasbourg, France